CLINICAL TRIAL: NCT07011888
Title: Current and Innovative Physiotherapy Practices in Stroke Rehabilitation: A Clinical Case Report
Brief Title: Innovative Physiotherapy in Stroke Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sevval Yesilkır (Other)
Responsible Party: Sponsor-Investigator, Sevval Yesilkır, Physiotherapist, MSc, Medipol University
Organization: Medipol University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3288; E-10840098-202.3.02-3288 (Registry Identifier: Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic; Chronic Stroke Survivors
Keywords: chronic stroke; Saebo; ultrasound therapy; vestibular training; stroke rehabilitation; balance; case report; functional independence
MeSH Terms: conditions — Ischemic Stroke | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-group interventional study involving one participant who will receive a rehabilitation program including VRT, ultrasound therapy, NMES, and the use of SaeboStim GO and Saebo Glove devices. The study aims to evaluate the effects of this combined intervention on motor skills, balance, gait ability, independence in daily activities, and cognitive functions over the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single-Case Rehabilitation Intervention (Experimental): This arm involves a rehabilitation program for a chronic stroke patient including VRT (Vestibular Rehabilitation Therapy), therapeutic ultrasound, and use of SaeboStim GO device combined with Saebo Glove orthosis to improve motor skills, balance, gait, activities of daily living, and cognitive functions.
  Interventions: Device: SaeboStim GO with Saebo Glove Rehabilitation Program

INTERVENTIONS:
Device: SaeboStim GO with Saebo Glove Rehabilitation Program — The intervention consists of a comprehensive rehabilitation program for a chronic stroke patient, utilizing the SaeboStim GO device combined with the Saebo Glove orthosis to facilitate and strengthen hand and upper limb motor function. The program also includes therapeutic ultrasound to support tissue healing, and vestibular rehabilitation therapy (VRT) to enhance motor learning and engagement. This combined approach aims to improve motor skills, balance, gait, daily living activities, and cognitive functions over a treatment period of six months.
  Other Names: vestibular rehabilitation therapy; therapeutic ultrasound

SUMMARY:
This study reports a single-case rehabilitation program for a chronic stroke patient focusing on innovative physiotherapy techniques. Over six weeks, the patient will undergo combined treatments including vestibular rehabilitation therapy, ultrasound therapy, and functional hand therapy using Saebo devices. The goal is to improve motor functions and daily living independence. This report aims to share clinical insights and outcomes to support stroke rehabilitation practices.

DETAILED DESCRIPTION:
This single-case clinical report presents a comprehensive rehabilitation program for a stroke patient over a period of six weeks. The intervention consists of three main components:

1. Vestibular Rehabilitation Therapy (VRT): Exercises aimed at improving ocular motor control, balance, and vestibulo-ocular reflex through specific eye movements and walking patterns, progressing in difficulty over time.
2. Ultrasound Therapy: Application of low-frequency portable ultrasound to targeted muscle groups to reduce spasticity and promote muscle relaxation, performed in prone or side-lying positions.
3. Functional Hand Rehabilitation: Use of SaeboStim GO and Saebo Glove devices to reduce spasticity in upper limb muscles and enhance hand function through electrical stimulation and active-assisted exercises.

Throughout the program, treatment sessions are conducted three times weekly, each lasting two hours. Outcomes related to motor improvement, spasticity reduction, and functional independence are monitored and evaluated using descriptive statistics and time-series analysis.

The purpose of this report is to provide detailed clinical insights into the application of combined innovative physiotherapy methods in stroke rehabilitation and to highlight their potential benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosis of chronic ischemic stroke (more than 6 months post-stroke).
* Presence of motor dysfunction, balance impairment, or gait difficulties related to stroke.
* Willingness and ability to participate in a comprehensive rehabilitation program involving physical therapy and device-assisted interventions (e.g., SaeboStim GO, Saebo Glove).

Exclusion Criteria:

* Presence of uncontrolled systemic diseases or active infections that would interfere with rehabilitation.
* Severe psychiatric disorders that would impede participation.
* Contraindications to the use of physical therapy devices or interventions used in the study.
* Severe orthopedic conditions that preclude participation in the rehabilitation program.

Ages: 50 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | The beginning of study and after 6 weeks
  The Barthel Index (BI) is a widely used functional assessment tool developed to assess an individual's level of independence in activities of daily living. It assesses ten basic categories, including feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfers (bed to chair), mobility on flat surfaces, and stair climbing. Each category is scored based on the level of assistance the individual requires; the total scores ranges from 0 to 100, with higher scores indicating greater functional independence. Score between 0-20 indicate severe dependency, 21-60 moderate dependency, 61-90 mild dependency, 91-99 near-complete independence, 100 complete independence. The Turkish version of the Barthel Index has been validated for clinical use.
The Montreal Cognitive Assessment | The beginning of study and after 6 weeks
  The Montreal Cognitive Assessment (MoCA) is a short, multidimensional cognitive assessment tool developed to detect mild cognitive impairments in the early stages. The test aims to measure performance in various cognitive domains such as attention and concentration, executive functions, memory, language, visual-spatial skills, abstraction, calculation, and orientation in time and space. The MoCA is scored out of a total of 30 points, and based on generally accepted thresholds, a score of 26 and above indicates normal cognitive functioning, while a score of 25 and below indicates a risk of cognitive impairment. Since educational level may affect the result, it is recommended to add one point to the final score for individuals with less than 12 years of education. A validated Turkish version of the MoCA is used in this study.
Modified Falls Efficacy Scale | The beginning of study and after 6 weeks
  The Modified Falls Efficacy Scale (MFES) is a self-report-based tool that assesses the fear of falling individuals experience while performing their daily activities. The scale consists of 14 items, each scored between 0 (no confidence) to 10 (complete confidence). The highest possible total score is 140, with an average score of up to 10. Higher average scores indicate a low fear of falling during the activity, while lower scores indicate a high level of fear. The Turkish version of the MFES has been validated for use in clinical assessments.
Fugl-Meyer Assessment | The beginning of study and after 6 weeks
  Fugl-Meyer Assessment (FMA) originally evaluates five components: lower extremity motor function (FMA-LE, maximum score 34) and upper extremity motor function (FMA-UE, maximum score 66), sensory function (maximum score 24), balance (maximum score 14), range of motion (maximum score 44) and joint pain (maximum score 44). Two areas will be evaluated in this study: FMA-LE and FMA-UE. FMA-LE includes six categories such as basic reflex movements in the lower extremity, voluntary movements with muscle synergies, coordination and movement speed (tremor, dysmetria, timing). Most tasks are scored between 0 and 2; 0 indicates no movement, 1 partial movement and 2 correct movement. The FMA-UE assesses nine categories for the upper extremity: primary reflexes, flexor synergy, extensor synergy, combined synergy movements, out-of-synergy movements, wrist movements, hand movements, and coordination (tremor, dysmetria, speed). Most tasks are similarly scored from 0 to 2.
Wolf Motor Function Test | The beginning of study and after 6 weeks
  The Wolf Motor Function Test (WMFT) is a timed-based, task-oriented performance test developed to assess upper extremity motor function following stroke. This test, which consists of 15 tasks in total, allows for the monitoring of changes in motor skills over time. The first six tasks involve timed movements of joint segments, while the remaining nine tasks evaluate holistic functional movements. Each task is scored both for completion time (in seconds) and movement quality on a scale from 0 to 5 with the maximum score is 75. The WMFT provides both qualitative and quantitative data, making it a reliable tool for tracking rehabilitation progress.
Berg Balance Scale | The beginning of study and after 6 weeks
  The Berg Balance Scale (BBS) is a highly clinically valid and reliable tool used to assess balance performance. It is especially preferred for older adults and individuals with neurological disorders such as stroke, to determine the risk of falling due to balance issues. The scale consists of 14 tasks, each scored from 0 to 4, with a maximum total score of 56. The tasks include sitting, standing, turning, bending, and standing on one leg, covering a range of functional balance abilities. Lower scores are associated with a higher risk of falling; scores below 45 are generally considered clinically significant for fall risk.
Timed Up and Go Test | The beginning of study and after 6 weeks
  The Timed Up and Go Test (TUG) is a time-based test used to measure functional mobility and fall risk by assessing how long it takes for an individual to complete a sequence of daily movements. It is frequently used to objectively assess mobility levels in older adults and patients with neurological or orthopedic conditions. During the test, the individual rises from the chair, walks three meters forward, turns around, walks back to the starting point, and sits down again. This process is timed in seconds using a stopwatch. Times under 10 seconds are considered normal levels of mobility; values between 11 and 14 seconds indicate mild mobility limitation; times over 15 seconds are associated with reduced functional independence and increased fall risk. Times above 20 seconds may raise concerns about the ability to live independently; and times exceeding 30 seconds indicate severe mobility impairment and a high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Sevval Yesilkır, MSc, Principal Investigator; Gizem Ergezen Sahin, Dr. Assistant Professor, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study involves a single patient case report, and sharing individual participant data may compromise patient privacy and confidentiality. Therefore, IPD sharing is not planned.